CLINICAL TRIAL: NCT01418677
Title: An Open-Label Phase 1 Study to Assess the Pharmacokinetics and Safety of HALAVEN in Subjects With Cancer Who Also Have Impaired Renal Function
Brief Title: An Open-Label Study to Assess the Pharmacokinetics and Safety of HALAVEN in Subjects With Cancer Who Also Have Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7389-A001-106
Record Dates: First submitted 2011-08-01; First posted 2011-08-17 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: Unspecified Advance Solid Tumor, Protocol Specific
MeSH Terms: interventions — eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Active Comparator)
  Interventions: Drug: E7389
- Cohort 2 (Active Comparator)
  Interventions: Drug: E7389
- Cohort 3 (Active Comparator)
  Interventions: Drug: E7389

INTERVENTIONS:
Drug: E7389 — Severe renal impairment-the dose to be administered will be based on the interim analyses of safety and pharmacokinetics in subjects with moderate renal impairment (Cohort 1).
  Other Names: Halaven
  Arms: Cohort 1
Drug: E7389 — Moderate renal impairment-HALAVEN will be dosed at 1.4 mg/m2.
  Other Names: Halaven
  Arms: Cohort 2
Drug: E7389 — Normal renal function-HALAVEN will be dosed at 1.4 mg/m2.
  Other Names: Halaven
  Arms: Cohort 3

SUMMARY:
This is an open-label non-randomized study in subjects with advanced or metastatic solid tumors who are no longer responding to available therapy. HALAVEN will be administered to subjects on Days 1 and 8 of a 21-day cycle.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced solid tumors that have progressed following standard therapy or for which no standard therapy exists (including surgery or radiation therapy).
* Renal function must fall into one of the following categories:
* Normal function - creatinine clearance greater than or equal to 80 mL/min.
* Moderate impairment - creatinine clearance >30 to 50 mL/min.
* Severe impairment - creatinine clearance 15 to less than 30 mL/min.
* Adequate liver function as evidenced by bilirubin less than or equal to 1.5 times the upper limit of normal (ULN) and alkaline phosphatase (ALP), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) less than or equal to 3 times the ULN (in the case of liver metastasis less than or equal to 5 times ULN). In the case ALP >3 times the ULN (in the absence of liver metastasis) or >5 times the ULN (in the presence of liver metastasis), and the subject is also known to have bone metastasis, the liver specific ALP must be separated from the total and used to assess the liver function instead of the total ALP.

Exclusion Criteria:

* Subjects with mild renal impairment (creatinine clearance greater than 50 to less than 80 mL/min).
* Subjects with end stage renal disease (creatinine clearance less than 15 mL/min or on dialysis).
* Subjects with a hypersensitivity to halichondrin B and/or halichondrin B chemical derivatives.
* Subjects with prior participation in an HALAVEN clinical study, even if not previously assigned to HALAVEN treatment.
* Radiation therapy encompassing >30 % of bone marrow.
* Subjects with organ allografts requiring immunosuppression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-10; Primary Completion 2014-07 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
To study the influence of moderate and severe renal impairment on the Composite of Pharmacokinetics of HALAVEN following a single intravenous administration to subjects with cancer. | Halaven will be measured on Day 1 and 8 of a 21 day cycle.
  The primary analysis will be conducted using the dose-normalized primary PK parameters (AUC0-inf, AUC0-last, and Cmax) respectively. Relationships between each individual PK parameter and renal function (creatinine clearance) will be analyzed by linear regression models using the PK parameter as the dependent variable and renal function as the independent variable.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability of HALAVEN in subjects with moderate or severe renal impairment, as well as in those with normal renal function. | Halaven will be measured on Day 1 and 8 of a 21 day cycle.
  Safety data that will be evaluated include adverse events, clinical laboratory results, physical examination results, ECG, and vital signs

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Duarte, California
  - Miami, Florida
  - Atlanta, Georgia
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - New Brunswick, New Jersey
  - The Bronx, New York
  - San Antonio, Texas

REFERENCES:
- [Derived] Tan AR, Sarantopoulos J, Lee L, Reyderman L, He Y, Olivo M, Goel S. Pharmacokinetics of eribulin mesylate in cancer patients with normal and impaired renal function. Cancer Chemother Pharmacol. 2015 Nov;76(5):1051-61. doi: 10.1007/s00280-015-2878-5. Epub 2015 Oct 3. PMID 26433580